CLINICAL TRIAL: NCT07313865
Title: From Commensalism to Pathogenicity: Exploring the Pathophysiology of Bacteremia to Better Understand Enterococcus Faecalis Infective Endocarditisléter
Brief Title: From Commensalism to Pathogenicity: Exploring the Pathophysiology of Bacteremia to Better Understand Enterococcus Faecalis Infective Endocarditis
Acronym: BAC-ENDO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RBHP 2025 VIDAL
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Infective Endocarditis (IE)
Keywords: Enterococcus faecalis; Bacteremia; Dysbiosis; Pathophysiology; Virulence factors
MeSH Terms: conditions — Endocarditis; Bacteremia; Dysbiosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cases (Other): Collection of four swabs (two rectal swabs, one oral swab, and one skin swab from the inguinal fold).
  Interventions: Biological: Microbiological sampling (swab collection)
- Controls (Other): Collection of a single rectal swab.
  Interventions: Biological: Microbiological sampling (swab collection)

INTERVENTIONS:
Biological: Microbiological sampling (swab collection) — Participants in the case group will undergo microbiological sampling consisting of four swabs: two rectal swabs, one oral swab, and one skin swab from the inguinal fold.
  Participants in the control group will undergo a single rectal swab. The samples will be collected for microbiological analysis.

SUMMARY:
Enterococci are pathobionts of the human intestinal microbiota: they colonize the gastrointestinal tract as well as the skin, urine, wounds, bile, the oral cavity and endodontic canal, and medical devices (urinary catheters, venous catheters, etc.). They are responsible for urinary, dental, bloodstream, endocardial, biliary, and gastrointestinal infections.

Enterococcus faecalis is the enterococcus most frequently isolated from clinical specimens. It is the third leading cause of infective endocarditis (infection of the cardiac valves) and the leading cause of endocarditis following TAVI (transcatheter aortic valve implantation via the femoral route). E. faecalis infective endocarditis (EFIE) is severe and difficult to treat, with a particularly high relapse rate despite appropriate antibiotic therapy.

Cardiac valve contamination is always secondary to E. faecalis bacteremia, particularly in cases of isolated E. faecalis bacteremia (EFIB), defined by the absence of an identifiable portal of entry. Once in the bloodstream, the bacterium adheres to the valvular endothelium (healthy or damaged) through specific virulence factors, including endocarditis- and biofilm-associated pili (ebp), the collagen adhesin Ace, and aggregation substance (Agg).

The classical portals of entry for EFIE are infections of the urinary tract and the gastrointestinal tract. However, despite extensive investigations, the source of infection remains unidentified in more than 50% of cases. An imbalance of the intestinal microbiota, leading to overgrowth and subsequent translocation of E. faecalis from the digestive tract into the bloodstream, could explain the absence of an identifiable portal of entry during routine clinical and paraclinical evaluations. This plausible hypothesis remains largely unexplored to date. A better understanding of the underlying pathophysiology-particularly gut dysbiosis and the pathogen's capacity for intestinal translocation-could improve the prevention of EFIE occurrence and relapse.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older;
* Capable of giving informed consent;
* Affiliated with a social security system;
* Hospitalized with at least one positive blood culture for Enterococcus faecalis, without an obvious clinical entry point after physical examination and initial routine investigations (BIEF group);
* Hospitalized for another bacteremia, without an obvious clinical entry point after initial routine investigations (Control group);
* Receiving antibiotic therapy that was started less than 48 hours ago

Exclusion Criteria:

* Refusal to participate in the study;
* Pregnant or breastfeeding women;
* Individuals under guardianship, curatorship, deprived of liberty, or under judicial protection;
* Antibiotic therapy for the current infectious episode started more than 48 hours prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Qualitative and quantitative bacterial composition of the intestinal microbiota (molecular microbiology/PCR). | From enrollment to the collection of the four swabs: 24 to 48 hours.

SECONDARY OUTCOMES:
Mapping of E. faecalis colonization (urinary, digestive, and/or cutaneous) in patients diagnosed with E. faecalis bacteremia (EFIB); | From enrollment to the collection of the four swabs: 24 to 48 hours.
Genomic characterization through core genome analysis of E. faecalis strains isolated from colonization sites and from blood cultures in the same patient diagnosed with EFIB; | From enrollment to the collection of the four swabs: 24 to 48 hours.
Whole-genome characterization of E. faecalis strains isolated from colonization sites and those recovered from blood cultures in patients with EFIB; | From enrollment to the collection of the four swabs: 24 to 48 hours.
Description of potential portals of entry for enterococci at the end of hospitalization for EFIB. | From enrollment to the collection of the four swabs: 24 to 48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Magali VIDAL, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France, France